CLINICAL TRIAL: NCT05112146
Title: Effects of Whey Protein Pre-meals on Post-prandial Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18.08BIO
Record Dates: First submitted 2021-09-30; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-09

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control 10 (Placebo Comparator): 100 ml Water taken 10 min before standard meal
  Interventions: Dietary Supplement: Water
- Whey protein isolate 10 (Experimental): 10 g whey protein isolate diluted in 100 ml taken 10 min before standard meal
  Interventions: Dietary Supplement: Whey protein isolate
- Whey protein microgel 10 (Experimental): 10g whey protein microgel in 100 ml taken 10 min before standard meal
  Interventions: Dietary Supplement: Whey protein microgel
- Control 30 (Placebo Comparator): 100 ml Water taken 30 min before standard meal
  Interventions: Dietary Supplement: Water
- Whey protein isolate 30 (Experimental): 10 g whey protein isolate diluted in 100 ml taken 30 min before standard meal
  Interventions: Dietary Supplement: Whey protein isolate
- Whey protein microgel 30 (Experimental): 10g whey protein microgel in 100 ml taken 30 min before standard meal
  Interventions: Dietary Supplement: Whey protein microgel

INTERVENTIONS:
Dietary Supplement: Whey protein isolate — Oral administration
  Arms: Whey protein isolate 10; Whey protein isolate 30
Dietary Supplement: Whey protein microgel — Oral administration
  Arms: Whey protein microgel 10; Whey protein microgel 30
Dietary Supplement: Water — Oral administration
  Arms: Control 10; Control 30

SUMMARY:
The aim of this project was to determine if an administration of either 10 g of whey protein isolate or 10 g of whey protein microgels 30 or 10 min before a standard meal could reduce postprandial glucose response in obese subjects.

DETAILED DESCRIPTION:
Monocentric, controlled, randomized, open, complete cross-over study design where participants will take 2 test products or water (negative control) at 2 different time points.

The targeted population will be 16 completely healthy males and females at risk for pre-diabetes.

Primary objective: To quantify the effects of whey protein pre-meals administrated at 30 or 10 min before a meal on post-prandial glucose in the interstitial tissue, as compared to water as negative control.

Secondary objective: To compare glucose response of the different pre-meals (water, whey protein isolate, whey protein micelles).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participant
* Age between 40 and 65 years
* BMI higher than 27.0 kg/m2
* Sedentarity (no more than 30 min of walk per day).
* Able to understand and sign an informed consent form

Exclusion Criteria:

* Any known metabolic disease including diabetes or chronic drug intake (aspirin, vitamin C and mineral supplements, steroids, protease inhibitors, antidepressants, anxiolytic, or antipsychotics…) possibly impacting (to the opinion of the medical doctor):
* The digestion or absorption of nutrients
* The postprandial glucose response
* Major medical/surgical event requiring hospitalization in the last 3 months, to the opinion of the medical doctor
* Known allergy and intolerance to products components
* Medically known cutaneous hypersensitivity to adhesives and plasters
* Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer.
* Smokers
* Volunteer who cannot be expected to comply with the protocol
* Subject having a hierarchical link with the research team members

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Post-prandial glucose | Hour 0 to hour 2 after standard meal consumption
  Incremental area under the curve

SECONDARY OUTCOMES:
C max glucose | Hour 0 to hour 2 after standard meal consumption
  Incremental Cmax
T max glucose | Hour 0 to hour 2 after standard meal consumption
  Incremental Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Christian Darimont, Principal Investigator — Nestlé Research
Locations (1):
- Nestlé Clinical Research Unit, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided